CLINICAL TRIAL: NCT06000865
Title: The GRADE Randomized Trial: Glaucoma Rehabilitation With Action viDeo Games and Exercise
Brief Title: Glaucoma Rehabilitation With Action viDeo Games and Exercise - GRADE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: University of Waterloo (Other); The University of Hong Kong (Other); University of Leicester (Other)
Responsible Party: Principal Investigator, Allen MY Cheong, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 15602821
Record Dates: First submitted 2022-09-25; First posted 2023-08-21 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-03

CONDITIONS: Glaucoma; Visual Impairment
Keywords: Glaucoma; Peripheral field loss; Action video games; Balance functions; Fear of falling; Quality of life
MeSH Terms: conditions — Glaucoma; Vision Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interactive action video-game training (AVG) (Active Comparator): AVG using a Nintendo Switch gaming station will be administered in 20 sessions over 10 weeks (45 minutes per session, 2 sessions per week). Participants will be in standing position with game controllers or sensors attached to the body while playing games involving muscle stretching and strengthening exercises.
  Interventions: Behavioral: Action video game training
- Conventional physical training (PT) (Experimental): Participants in the PT will receive 45-minutes conventional physical training.
  Interventions: Behavioral: Conventional physical training

INTERVENTIONS:
Behavioral: Action video game training — 20 sessions of AVG over 10 weeks (45 minutes per session, 2 sessions per week)
  Arms: Interactive action video-game training (AVG)
Behavioral: Conventional physical training — 20 sessions of physical training over 10 weeks (45 minutes per session, 2 sessions per week)
  Arms: Conventional physical training (PT)

SUMMARY:
Falls are one of the most serious public health concerns for seniors, with significant medical and economic consequences. This concern is even higher in patients with peripheral field loss due to glaucoma because of the patients' compromised visual input. The investigators' project proposes an innovative, entertaining, easily accessible and enjoyable intervention for improving mobility and postural control function in glaucoma patients with peripheral vision loss, who are more prone to falls and suffer from fear of falling. The new intervention examined in this project can be implemented in current vision and balance rehabilitation programs, and may benefit patients with different types of visual impairment to minimize their risk of falls and improve their quality of life.

DETAILED DESCRIPTION:
A prospective, 2-arm, randomized, single-blind, active-control trial will enroll 56 moderately- to severely-affected glaucoma patients with stable peripheral field loss, intact cognitive function, and no history of balance training. Participants will be randomly assigned 1:1 to one of two groups: 1) standing, physically interactive action video-game training (AVG_PI); and 2) conventional physical training (PT). AVG using a Nintendo Switch gaming station will be administered in 20 sessions over 10 weeks (45 minutes per session, 2 sessions per week). Participants in the AVG_PI will be in standing position with game controllers or sensors attached to the body while playing games involving muscle stretching and strengthening exercises. Participants in the PT will receive 45-minutes conventional physical training. Outcome measures will be assessed before training, and after 10 and 20 training sessions. The primary outcome measure is a test of mobility, and the secondary outcome measures include tests for dynamic balance plus visual cognition, static balance, visual cognition, and patient reported outcomes for fear of falling and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of moderate to severe bilateral glaucomatous optic neuropathy (GON) from primary open-angle (including normal tension) or angle-closure glaucoma, as determined by an ophthalmologist, with abnormal Glaucoma Hemifield Test on standard Humphrey Field Analyzer 24-2 testing and matching nerve-fiber layer thinning on optical coherence tomography;
2. Stable vision and visual field loss for at least 3 months;
3. With a best-corrected distance acuity of 6/12 or better (equivalent to 0.3 logMAR acuity or better to confirm that participant's central vision is preserved);
4. With a cognitive functional score of 22 or above in the Montreal Cognitive Assessment - Hong Kong version (to confirm participants' intact cognitive function).

Exclusion Criteria:

1. Advanced glaucoma with GON of median deviation worse than -25 decibel;
2. Ocular diseases other than glaucoma (e.g., age-related macular degeneration, diabetic retinopathy, and moderate to severe cataract);
3. Severe medical problems (e.g., stroke, Parkinson's disease) or self-reported neurological (e.g. brain surgery, brain tumor and peripheral neuropathy), or cognitive disorders (e.g., diagnosed dementia or cognitive impairment);
4. Physical impairments (e.g. need the use of orthopedic and mobility aids) or physical limitations restricting them from independent walking;
5. Self-reported or medically diagnosed vestibular/ cerebellar dysfunction, history of vertigo, or severe hearing loss;
6. Using any medications for any neurological conditions or psychiatric drugs (e.g. sedative, hypnotic) that might interfere motor control; and
7. Currently attending any intensive physical/balance training.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-09-09 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Gait Measure - Time Up and Go test combining Narrow path walking test | Change from baseline at week 5 and change from baseline at week 10.
  Time Up and Go test combining Narrow path walking test: All participants need to stand up from a 46 cm height chair, walk on the path at their usual pace until the strip of a non-reflective tape, cross over the tape, turn 180°, walk to the starting position and finally sit down. Then repeat the same procedure within a narrower width. Participants need to use the dominant leg to step onto the standing position on one force plate while the non-dominant leg stands on the other force plate.
  The test will repeat for 10 times. Participants' gait parameters including hip flexion/extension (degree), knee Min/Max (degree), ankle flexion/extension (degree), walking speed (mm/s), step width (mm), and step length(mm) will be measured and analyzed for each condition.

SECONDARY OUTCOMES:
Static Balance Measure | Change from baseline at week 5 and change from baseline at week 10.
  Static Balance: Participants will be asked to stand on a force place with a foam while performing visual searching. Parameters including maximum antero-posterior amplitude (mm), maximum medio-lateral amplitude (mm), total sway path (mm), and root mean square sway (mm/s) will be analyzed.
  Each test would be repeated for 3 times.
Perturbed Balance Measure | Change from baseline at week 5 and change from baseline at week 10.
  Perturbed Balance: Participants will be asked to stand on a force place which will translate forward or backward while performing visual searching. Parameters including latency (ms) reacting to the perturbation, maximum antero-posterior amplitude (mm), maximum medio-lateral amplitude (mm), total sway path (mm), and root mean square sway (mm/s) will be analyzed.
  Each test would be repeated for 3 times.
Useful field of view (UFOV) | Change from baseline at week 5 and change from baseline at week 10.
  Visual attention will be examined by Useful Field of View (UFOV). Participants will be asked to complete the following 3 tasks.
  1. Processing speed: Participants will be asked to discriminate the central presented stimulus as a target or distractor.
  2. Divided attention: In addition to discriminating the central target, participants are required to identify the location of the peripheral target.
  3. Selective attention: Procedure is similar as "Divided attention". Participants are required to identify the location of peripheral target among the distractors.
  Parameter includes time to reach threshold(ms)
Reaction time (RT) | Change from baseline at week 5 and change from baseline at week 10.
  Each participant is asked to complete the following task using a customized computer programme.
  Reaction Time Test: Participants will be asked to respond as fast as possible when the same stimulus (an 'x' emerging in a square in the middle of the screen) was presented.
  This test will be repeated for 3 blocks with 46 trials per block. Parameter includes reaction time to correct answer(ms).
Cognitive Reflection Test | Change from baseline at week 5 and change from baseline at week 10.
  Each participant is asked to complete the following task using a customized computer programme.
  Cognitive Reflection Test: Participants will be presented with four squares horizontally on the screen. They will be asked to react to an 'x' emerging in one of the squares (40 trials in total) by pressing a corresponding key on a keyboard-'1', '2', '3', or '4' which present the position of 'x' . Parameter includes reaction time to correct answer(ms).
Quality of Life Questionnaire measure | Change from baseline at week 5 and change from baseline at week 10.
  The effect of intervention on quality of life will be evaluated using the Learning Vector Quantization (LvQ) Scale.
  In the LvQ, participants will be asked to rate how much their eyesight has interfered with each of 24 activities in the past month. The completion results in a summed score between 0 (a low quality of life) and 125 (a high quality of life).
Fear of Falling Questionnaire measure | Change from baseline at week 5 and change from baseline at week 10.
  The effect of intervention on fear of falling will be evaluated using the Chinese versions of Falls Efficacy Scale International (FES-I).
  In the FES-I, participants will be asked "how concerned they are about the possibility of falling" for each of the 16 social and physical activities. The completion results in a summed score between minimum 16 (no concern about falling) to maximum 64 (severe concern about falling).

CONTACTS AND LOCATIONS:
Overall Officials: Allen Cheong, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication will be available upon reasonable request to the research team.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: IPD will be available no later than 6 months following publication and for 1 year.
Access Criteria: IPD will be shared with investigators who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Yihong P, Thompson B, Winser S, Lau I, Suen V, Cheung M, Cheong AMY. Glaucoma rehabilitation with action video games and exercise: study protocol of an active-controlled trial (GRADE). BMJ Open. 2025 Sep 17;15(9):e105971. doi: 10.1136/bmjopen-2025-105971. PMID 40967649